CLINICAL TRIAL: NCT00733954
Title: A Comparison Between Clobetasol Propionate (Clobex®) Spray and Clobetasol Propionate Ointment With Regard to Efficacy, Safety, Subject Satisfaction and Duration of Response in Moderate to Severe Plaque Psoriasis
Brief Title: Efficacy/Safety/Subject Satisfaction/Duration of Response of Clobetasol Propionate Spray vs Ointment in Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: US10012
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Results first posted 2009-08-20 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2014-04

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- clobetasol propionate spray (Active Comparator): clobetasol propionate spray 0.05%
  Interventions: Drug: clobetasol propionate spray
- clobetasol propionate ointment (Active Comparator): clobetasol propionate ointment 0.05%
  Interventions: Drug: clobetasol propionate ointment

INTERVENTIONS:
Drug: clobetasol propionate spray — Apply twice daily
  Other Names: Clobex® Spray
  Arms: clobetasol propionate spray
Drug: clobetasol propionate ointment — Apply twice daily
  Arms: clobetasol propionate ointment

SUMMARY:
This study is a comparison between Clobetasol Propionate Spray and Clobetasol Propionate Ointment with Regard to Efficacy, Safety, Subject Satisfaction and Duration of Response in Moderate to Severe Stable Plaque Psoriasis. Subjects will be enrolled and randomized into one of two groups: clobetasol propionate Spray for 4 weeks of treatment or clobetasol propionate ointment for 2 weeks of treatment with a 2 week follow-up visit for each group.

DETAILED DESCRIPTION:
Same as above.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of moderate to severe plaque psoriasis, defined as 3% - 20% of the body surface area. For the purposes of study treatment, most areas will be treated with the exception of face, scalp, groin, axillae and other intertriginous areas
* Overall disease severity is at least 3 (moderate)

Exclusion Criteria:

* Subjects who have surface area involvement too large that would require more than 50 grams per week of clobetasol propionate spray or more than 50 grams per week of clobetasol propionate ointment
* Subjects whose psoriasis involves only the scalp, face or groin
* Subjects with non-plaque psoriasis or other related diseases not classified as plaque psoriasis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (6):
- United States (6):
  - East Bay Dermatology Medical Group, Inc., Fremont, California
  - Solano Clinical Research, Vallejo, California
  - Henry Ford Medical Center, Detroit, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Dermatology Associates of Rochester, Rochester, New York
  - Baylor Research Institute - Dermatology Research, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject was enrolled on August 22, 2007 and the last subject enrolled was February 20, 2008. Investigative sites were located at academic institutions and private physician offices.
Pre-assignment Details: The specified wash-out period up to baseline was 14 days (topical steroid containing medication and/or UVB treatment, Dovonex, anthralin and/or tar); and 4 weeks (systemic corticosteroids, biologics and/or PUVA treatment).
Period: Overall Study
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Started | 124 | 125
Completed | 116 | 123
Not Completed | 8 | 2
Not completed — Lost to Follow-up | 5 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment | Total
Number analyzed (Participants) | 124 | 125 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (14.0) | 50.2 (13.5) | 50.4 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 43 | 95
  Male | 72 | 82 | 154

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Clear/Almost Clear of Plaque Psoriasis From Baseline to End of Treatment Based on the Overall Disease Severity (ODS) Scale
Description: Success Rate on Overall Disease Severity (ODS) scale (Clear/Almost Clear, Mild, Moderate, Severe/Very Severe with Clear/Almost Clear being best and Severe/Very Severe being worst) from Baseline to End of Treatment (wk 4 - clobetasol propionate spray; wk 2 - clobetasol propionate ointment)
Time Frame: Baseline and Week 2 and Baseline and Week 4
Population: Intent-to-treat (ITT), Last observation carried forward (LOCF)
Measure: Number; unit: Participants
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
Participants | 62 | 44

2. Secondary Outcome: Number of Participants Who Are Clear/Almost Clear of Plaque Psoriasis From Baseline to After Two Weeks of Treatment Based on the Overall Disease Severity (ODS) Scale
Description: Success Rate on Overall Disease Severity (ODS) scale (Clear/Almost Clear, Mild, Moderate, Severe/Very Severe) with Clear/Almost Clear being best and Severe/Very Severe being worst from Baseline to after 2 weeks of treatment
Time Frame: Baseline and Week 2
Measure: Number; unit: Participants
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
Participants | 39 | 44

3. Secondary Outcome: Number of Participants Who Are Clear/Almost Clear of Plaque Psoriasis From Baseline to 2 Weeks Post Treatment Based on the Overall Disease Severity (ODS) Scale
Description: Success Rate on Overall Disease Severity scale (Clear/Almost Clear, Moderate, Severe/Very Severe) with Clear/Almost Clear being best and Severe/Very Severe being worst at 2 weeks post treatment (week 6 - clobetasol propionate spray and week 4 - clobetasol propionate ointment)
Time Frame: Baseline and Week 4 and Baseline and Week 6
Population: ITT, LOCF
Measure: Number; unit: Participants
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
Participants | 50 | 33

4. Secondary Outcome: Number of Participants With Decrease in Signs of Psoriasis (Erythema) From Baseline to After Two Weeks of Treatment
Description: Success Rate of decrease in Signs of Psoriasis (erythema) scale (Clear/Almost Clear, Mild, Moderate, Severe/Very Severe) with Clear/Almost clear being success and all others being failure from Baseline to after 2 weeks of treatment
Time Frame: Baseline and Week 2
Population: ITT, LOCF
Measure: Number; unit: Participants
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
Participants | 29 | 33

5. Secondary Outcome: Number of Participants With Decrease in Signs of Psoriasis (Scaling) From Baseline to After Two Weeks of Treatment
Description: Success Rate of decrease in Signs of Psoriasis (scaling) scale (Clear/Almost Clear, Mild, Moderate, Severe/Very Severe) with Clear/Almost clear being success and all others being failure from Baseline to after 2 weeks of treatment
Time Frame: Baseline and Week 2
Population: ITT, LOCF
Measure: Number; unit: Participants
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
Participants | 53 | 72

6. Secondary Outcome: Number of Participants With Decrease in Signs of Psoriasis (Plaque Elevation) From Baseline to After Two Weeks of Treatment
Description: Success Rate of decrease in Signs of Psoriasis (plaque elevation) scale (Clear/Almost Clear, Mild, Moderate, Severe/Very Severe) with Clear/Almost clear being success and all others being failure from Baseline to after 2 weeks of treatment
Time Frame: Baseline and Week 2
Population: ITT, LOCF
Measure: Number; unit: Participants
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
Participants | 48 | 52

7. Secondary Outcome: Number of Participants With Decrease in Signs of Psoriasis (Erythema) From Baseline to End of Treatment
Description: Success Rate on decrease in Signs of Psoriasis (erythema) scale (Clear/Almost Clear, Mild, Moderate, Severe/Very Severe) with Clear/Almost Clear being success and all others failure from Baseline to end of treatment (week 4 for clobetasol propionate spray and week 2 for clobetasol propionate ointment)
Time Frame: Baseline and Week 2 and Baseline and Week 4
Population: ITT, LOCF
Measure: Number; unit: Participants
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
Participants | 53 | 33

8. Secondary Outcome: Number of Participants With Decrease in Signs of Psoriasis (Scaling) From Baseline to End of Treatment
Description: Success Rate on decrease in Signs of Psoriasis (scaling) scale (Clear/Almost Clear, Mild, Moderate, Severe/Very Severe) with Clear/Almost Clear being success and all others being failure from Baseline to end of treatment (week 4 for clobetasol propionate spray and week 2 for clobetasol propionate ointment)
Time Frame: Baseline and Week 2 and Baseline and Week 4
Population: ITT, LOCF
Measure: Number; unit: Participants
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
Participants | 73 | 72

9. Secondary Outcome: Number of Participants With Decrease in Signs of Psoriasis (Plaque Elevation) From Baseline to End of Treatment
Description: Success Rate on decrease in Signs of Psoriasis (plaque elevation) scale (Clear/Almost Clear, Mild, Moderate, Severe/Very Severe) with Clear/Almost Clear being success and all others being failure from Baseline to end of treatment (week 4 for clobetasol propionate spray and week 2 for clobetasol propionate ointment)
Time Frame: Baseline and Week 2 and Baseline and Week 4
Population: ITT, LOCF
Measure: Number; unit: Participants
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
Participants | 72 | 52

10. Secondary Outcome: Number of Participants With Decrease in Signs of Psoriasis (Erythema) From Baseline to Two Weeks Post Treatment
Description: Success Rate on decrease in Signs of Psoriasis (erythema) scale (Clear/Almost Clear, Mild, Moderate, Severe/Very Severe) with Clear/Almost Clear being success and all others being failure from Baseline to 2 weeks post treatment (week 6 for clobetasol propionate spray and week 4 for clobetasol propionate ointment)
Time Frame: Baseline and Week 4 and Baseline and Week 6
Population: ITT, LOCF
Measure: Number; unit: Participants
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
Participants | 48 | 32

11. Secondary Outcome: Number of Participants With Decrease in Signs of Psoriasis (Scaling) From Baseline to Two Weeks Post Treatment
Description: Success Rate on decrease in Signs of Psoriasis (scaling) scale (Clear/Almost Clear, Mild, Moderate, Severe/Very Severe) with Clear/Almost Clear being success and all others being failure from Baseline to 2 weeks post treatment (week 6 for clobetasol propionate spray and week 4 for clobetasol propionate ointment)
Time Frame: Baseline and Week 4 and Baseline and Week 6
Population: ITT, LOCF
Measure: Number; unit: Participants
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
Participants | 56 | 43

12. Secondary Outcome: Number of Participants With Decrease in Signs of Psoriasis (Plaque Elevation) From Baseline to Two Weeks Post Treatment
Description: Success Rate on decrease in Signs of Psoriasis (plaque elevation) scale (Clear/Almost Clear, Mild, Moderate, Severe/Very Severe) with Clear/Almost Clear being success and all others being failure from Baseline and 2 weeks post treatment (week 6 for clobetasol propionate spray and week 4 for clobetasol propionate ointment)
Time Frame: Baseline and Week 4 and Baseline and Week 6
Population: ITT, LOCF
Measure: Number; unit: Participants
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
Participants | 55 | 35

13. Secondary Outcome: Percent Decrease in Body Surface Area Affected (%BSA Affected) From Baseline to After Two Weeks of Treatment
Description: Percent decrease in Body Surface Area affected (% BSA affected) from Baseline to after two weeks of treatment
Time Frame: Baseline and Week 2
Population: ITT, LOCF
Measure: Mean (Standard Deviation); unit: % BSA
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
% BSA | 28.6 (28) | 35.9 (30.5)

14. Secondary Outcome: Percent Decrease in Body Surface Area Treated (%BSA Treated) From Baseline to After Two Weeks of Treatment
Description: Percent decrease from baseline in Body Surface Area treated (% BSA treated) from Baseline to after two weeks of treatment
Time Frame: Baseline and Week 2
Population: ITT, LOCF
Measure: Mean (Standard Deviation); unit: % BSA
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
% BSA | 29.1 (29.6) | 38.4 (33.0)

15. Secondary Outcome: Percent Decrease in Body Surface Area Affected (%BSA Affected) From Baseline to End of Treatment
Description: Percent decrease in body surface area affected (%BSA affected) from Baseline to end of treatment (week 4 for clobetasol propionate spray and week 2 for clobetasol propionate ointment)
Time Frame: Baseline and Week 2 and Baseline and Week 4
Population: ITT, LOCF
Measure: Mean (Standard Deviation); unit: % BSA
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
% BSA | 51 (36.5) | 35.9 (30.5)

16. Secondary Outcome: Percent Decrease in Body Surface Area Treated (%BSA Treated) From Baseline to End of Treatment
Description: Percent decrease from baseline in body surface area treated (%BSA treated) from Baseline to end of treatment (week 4 for clobetasol propionate spray and week 2 for clobetasol propionate ointment)
Time Frame: Baseline and Week 2 and Baseline and Week 4
Population: ITT, LOCF
Measure: Mean (Standard Deviation); unit: % BSA
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
% BSA | 52 (37.5) | 38.4 (33.0)

17. Secondary Outcome: Percent Decrease in Body Surface Area Affected (%BSA Affected) From Baseline to Two Weeks Post Treatment
Description: Percent decrease in body surface area affected (%BSA affected) from Baseline two weeks post treatment (week 6 for clobetasol propionate spray and week 4 for clobetasol propionate ointment)
Time Frame: Baseline and Week 4 and Baseline and Week 6
Population: ITT, LOCF
Measure: Mean (Standard Deviation); unit: % BSA
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
% BSA | 48 (36.3) | 37.6 (34.4)

18. Secondary Outcome: Percent Decrease in Body Surface Area Treated (%BSA Treated) From Baseline to Two Weeks Post Treatment
Description: Percent decrease in body surface area treated (%BSA treated) from Baseline to two weeks post treatment (week 6 for clobetasol propionate spray and week 4 for clobetasol propionate ointment)
Time Frame: Baseline and Week 4 and Baseline and Week 6
Population: ITT, LOCF
Measure: Mean (Standard Deviation); unit: % BSA
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
% BSA | 48.6 (38.0) | 38.3 (37.9)

19. Secondary Outcome: Number of Participants With Tolerability Assessments Resulting in Adverse Events From Baseline to Two Weeks Post Treatment
Description: Number of Participants with Tolerability assessments (Pruritus, Telangiectasias, Stinging/Burning, Skin atrophy, Folliculitis) resulting in adverse events from Baseline to two weeks post treatment (week 6 for clobetasol propionate spray and week 4 for clobetasol propionate ointment)
Time Frame: Baseline and Week 4 and Baseline and Week 6
Population: Safety
Measure: Number; unit: Participants
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Number analyzed (Participants) | 124 | 125
Participants | 1 | 0

ADVERSE EVENTS:
Arm/Group | Clobetasol Propionate Spray | Clobetasol Propionate Ointment
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/123
Other Adverse Events (participants affected / at risk) | 0/122 | 0/123

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator has the right to publish or present the data results from this study, with agreed upon reviews by all interested parties, and in accordance with any confidentiality agreements that may exist.